CLINICAL TRIAL: NCT06919601
Title: Support Sessions for Parents With Children in the Pediatric Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-FY2022-338
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Parent Support
Keywords: parents grief intensive care support; death of child; death, grief, parent, child
MeSH Terms: conditions — Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Support Sessions for Parents on Expressing Grief (Experimental): Parents in the experiment group will receive 8 Grief-informed support sessions. Each session is curriculum driven and completed in a group session. each session lasts 1 hour. Each session will be delivered by a trained person in grief and loss.
  Interventions: Behavioral: Grief-Informed Healing Circles

INTERVENTIONS:
Behavioral: Grief-Informed Healing Circles — Eight one-hour sessions delivered in a group setting

SUMMARY:
The goal of this clinical trial is to learn if Grief-informed Parent Support sessions offered weekly to parents with a child in the pediatric intensive care unit work to decrease symptoms of parent grief compared to a non-grief informed parent support program offered weekly to parents with a child in the pediatric intensive care unit. The main question is:

Do parents with a child in the pediatric intensive care unit report fewer symptoms of grief, such as depression and anxiety, following their attendance at a parent support program with a grief-informed intervention compared to parents who receive a non-grief informed support program.

Participants will be randomized to :

Receive a 8-session grief-informed parent support program or a 8-session non grief-informed parent support program. Parents will report symptoms of grief before and after the 8-session parent support program.

DETAILED DESCRIPTION:
Grief is the response to a loss. Infants and children in intensive care units are at increased risk for chronic morbidity and death. Grief is a normal response to the potential or actual loss of a child. Grief related disorders of Post-Traumatic Stress Disorder (PTSD), anxiety, depression, and insomnia are reported by parents of children in PICU's.

To test the efficacy and impact of a grief-informed intervention, 100 parents of infants and children admitted to a PICU were recruited, within the first 7 days of admission. Fifty parents were randomized to 8, 1-hour grief informed sessions, led by a trained facilitator that followed a curriculum of validating grief and inviting each parent to share their grief.

Fifty parents were randomized to 8, 1-hr attention control sessions, led by a registered nurse, who offered guided imagery, meditation, and chair-based exercises. Attendance at sessions was recorded to establish dose and intervention efficacy. Following the 8 sessions, parents were administered the Parent Experiences Questionnaire (PEQ) to measure the 4 domains of: Unresolved Sorrow and Anger, Guilt and Worry, Long-Term Uncertainty, and Emotional Resources. Sixty-Four (64) parents completed the PEQ measure. Thirty-eight (38) of the 63 parents joined a second study to measure the PEQ four domains and parent and sibling behavioral functioning every 3 months for 12 months. A final qualitative interview will be offered to each parent completing the study (estimated 30 parents) and qualitative data triangulated with PEQ scores.

Attendance at the grief informed, Healing Circles Intervention, sessions was TWICE that of the attention control sessions. The differential scores of the four domains of the Parent Experiences Questionnaire were measured at 2 weeks after last session and at 3-, 6-, 9-, and 12 months. The PEQ four domain and total scores were correlated to Parent and Sibling functioning, as measured on the Adult and Child Behavior Checklist, respectively. Behavior functioning scores were scored as pre-clinical/clinical behaviors and non-clinical behaviors. All data was modeled to learn predictive patterns to best inform clinical practices for siblings and parents of children in the Pediatric Intensive Care Unit (PICU).

ELIGIBILITY:
Inclusion Criteria:

- Parent of a child in the pediatric intensive care unit

Exclusion Criteria:

- Not a parent of a child in the pediatric intensive care unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
parent grief | 12 months
  number of parent grief symptoms, such as depression and anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Judith M McFarlane, DrPH, Principal Investigator — Texas Woman's University
Locations (1):
- Texas Woman's University, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
outcome measure of parent grief and 8-session grief-informed intervention
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: June 2025 - December 2026
Access Criteria: From the investigator at jmcfarlane@twu.edu